CLINICAL TRIAL: NCT02287974
Title: Clinical Trial I/II Opened, Randomized and Controlled for the Study of the Use of Stem Cells Therapy in Insulinized Diabetic Patients Type 2 With Critical Ischemia in Lower Limbs: Study of the Needs of Insulin
Brief Title: Clinical Trial I/II Opened, Randomized and Controlled for the Study of the Use of Stem Cells Therapy in Insulinized Diabetic Patients Type 2 With Critical Ischemia in Lower Limbs (CLI): Study of the Needs of Insulin
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patients' numebr randomized not achieved. Investigators team with lack of interest and commitment. The sponsor closed prematurely patients' recruitment.
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CeTMMoTa/ICPDI/2010
Record Dates: First submitted 2013-02-25; First posted 2014-11-11 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-07

CONDITIONS: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Autologous mononuclear stem cell from the bone marrow (Experimental): Autologous mononuclear stem cell from the bone marrow in an unique infusion of 150-250 millions of cells
  Interventions: Drug: Stem cell infusion
- Autologous endothelial stem cell from the bone marrow (Experimental): Autologous endothelial progenitor CD133 stem cell from the bone marrow in an unique infusion of 2 - 7 millions of CD133 cells
  Interventions: Drug: Stem cell infusion
- Autologous mesenchymal stem cells from the adiposite tissue (Experimental): Autologous mesenchymal stem cells from the adipose tissue in an unique infusion of 0.5 millions of cells
  Interventions: Drug: Stem cell infusion
- Current medication for the disease (Active Comparator): Current medication for the disease
  Interventions: Drug: Stem cell infusion

INTERVENTIONS:
Drug: Stem cell infusion — Unique stem cell infusion of the randomized group

SUMMARY:
To study the effect of the stem cells therapy autologous mononuclear from the bone marrow, autologous progenitor endothelial CD133 cells from the bone marrow and autologous mesenchymal stem cells from adipose tissue on the inflammatory cytokines, the resistance to insulin and the decrease of the needs of insulin, besides evaluates the safety, viability and efficiency of the intra-arterial infusion of stem cells in diabetic patients type 2 with CLI.

DETAILED DESCRIPTION:
To study the effect of the stem cells therapy autologous mononuclear from the bone marrow, autologous progenitor endothelial CD133 cells from the bone marrow and autologous mesenchymal stem cells from adipose tissue on the inflammatory cytokines, the resistance to insulin and the decrease of the needs of insulin, besides evaluates the safety, viability and efficiency of the intra-arterial infusion of stem cells in diabetic patients type 2.

Diabetic patients will include with critical ischemia chronicle of at least a low member limb (CLI) and without possibilities of revascularization. 48 evaluable patients will be included, of which 36 patients will be included in the experimental group (12 for every cellular group) and 12 in the group control by conventional treatment. The population to studying will be constituted by 48 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤ 85 years
2. Diabetic type 2, in treatment with insulin at least 3 previous months.
3. Vascular disease infrapopliteal atherosclerotic of severe degree (Patients with category Rutherford-Becker ≥ 4), pretty or bilateral. The critical ischemia of the foot is defined as a persistent / persistent pain that needs analgesia and / or not healing present sores> 4 weeks, without evidence of improvement with conventional therapies and / or walking test between 1-6 minutes in two ergometries separated at least for 2 weeks and / or index ankle - arm in rest <0,8.
4. Impossibility of revascularization surgical or endovascular or I fail in the surgery of revascularization performed at least 30 days before, with persistence or entry in phase of critical ischemia
5. Life expectancy > 2 years.
6. Major amputation is not foreseen in any of the members in the next 6 months after the incorporation.
7. Normal Biochemical and bone marrow parameters defined for:

   * Leukocytes ≥ 3000
   * Neutrophils ≥ 1500
   * Platelets ≥ 140000
   * AST/ALT ≤ 2,5 standard range institution
   * Creatinine ≤2,5 mg/dl and explanation of creatinine ≤ 30 ml/min (MDRD4)
8. The women in fertile age will have to obtain negative results in a pregnancy test realized in the moment of the incorporation in the study and promise to use a contraceptive method medically approved while the study lasts.
9. Patients who give his Informed Consent in writing for the participation in the study. 10. Patients who have not taken part in another clinical trial in the last 3 months before the incorporation.

Exclusion Criteria:

1. Precedent of neoplasia or hematologic disease (disease myeloproliferative, syndrome myelodysplasic or leukaemia) in the last 2 years.
2. Major previous amputation.
3. Patients with arterial uncontrolled hypertension (defined as arterial tension> 180/110 in more than one occasion).
4. Cardiac severe insufficiency (NYHA the IVth) or Fraction of Ejection of left ventricle (FAITH) lower than 30 %.
5. Patients with ventricular malignant arrhythmias or unstable angina.
6. Diagnosis of venous deep thrombosis in 3 previous months.
7. Patients with genotype DD of the ECA or genotype E4 of the apo E.
8. Concomitant therapy that includes oxygen hyperbaric, vasoactive substances, agents against angiogenesis or inhibiting Cox-II. The agents use is allowed antiplatelets.
9. Index of corporal mass> 40 Kg/m2.
10. Patients with the diagnosis of alcoholism in the moment of the incorporation.
11. Proliferative Retinopathy without possibility of treatment.
12. Diabetic Nephropathy with haemodialysis
13. Concomitant disease that reduces the life expectancy to less than 1 years.
14. Impossibility foreseen to obtain the inhaled one of 100ml of bone marrow.
15. Infection for HIV, Hepatitis B or Hepatitis C.
16. Impede in the follow-up.
17. ACV or heart attack of myocardium in the last 3 months
18. Anaemia (Haemoglobin <7.9 g/dl)
19. Patients before treated with cellular therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | the entire follow-up period, in the first 24 hours after the infusion of stem cells
  To evaluate the possible complications derived from the procedure (in the first 24 hours after the infusion of stem cells and the incident of Serious Adverse Events and not Serious Adverse Events related to the IMPD or to the procedure of administration

SECONDARY OUTCOMES:
Efficacy measured by: The changes in the requirements of insulin, Peptide C, Resistance to the insulin, inflammatory Cytokines, pancreatic Reservation, Quantification of the degree of neovascularization (angio/arteriogenesis and vasculogenesis) | 6 months
  Efficacy measured by: The changes in the requirements of insulin, Peptide C, Resistance to the insulin, inflammatory Cytokines, pancreatic Reservation, Quantification of the degree of neovascularization (angio/arteriogenesis and vasculogenesis) after 6 months of the stem cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bernat Soria, Principal Investigator — CABIMER (Centro Andaluz de Biología Molecular y Medicina Regenerativa)
Locations (2):
- Spain (2):
  - Hopsital U. Virgen Macarena, Seville, Seville
  - CABIMER (Andalusian Center for Molecular Biology and Regenerative Medicine), Seville